CLINICAL TRIAL: NCT05638425
Title: An Observational Study on the Efficacy and Safety of Radiotherapy Combined With PD-1 Inhibitors and Chemotherapy in the Treatment of NSCLC Patients With Symptomatic Brain Metastases
Brief Title: Radiotherapy Combined With PD-1 Inhibitors and Chemotherapy in the Treatment of NSCLC Patients With Symptomatic Brain Metastases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ESRCPIC
Record Dates: First submitted 2022-11-27; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Brain Metastases
Keywords: radiotherapy; PD-1; symptomatic brain metastases; non-small cell lung cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Radiation: Radiotherapy combined with PD-1 inhibitors

INTERVENTIONS:
Radiation: Radiotherapy combined with PD-1 inhibitors — Radiotherapy should be carried out within 4 weeks after the first dose of PD-1 inhibitor; the radiotherapy method should be determined according to the patient's condition; PD-1 inhibitor and chemotherapy should refer to the actual product instructions

SUMMARY:
This is a prospective, single-center observational clinical study aimed at the efficacy and safety of radiotherapy combined with PD-1 inhibitors and chemotherapy in the treatment of Chinese patients with symptomatic NSCLC with brain metastases.

DETAILED DESCRIPTION:
Radiotherapy is carried out within 4 weeks after the first dose of PD-1 inhibitor; radiotherapy is determined according to the patient's condition; the use of PD-1 inhibitors and chemotherapy is based on the actual product instructions.

From December 2021 to December 2023, after the patients signed the informed consent, they will be included in this observational study after being assessed as meeting the inclusion criteria. A total of 20 cases are planned to be included for research analysis. All eligible patients meeting the inclusion and exclusion criteria will be invited to participate in this study. Patients included in the study will be solicited to allow efficacy evaluation and survival follow-up during the study and after treatment. Patients were considered to be on study unless the patient died, was withdrawn from the study, was lost to follow-up, or the study was terminated. Patients do not need to visit a doctor or receive evaluation specifically because of the study, and the study doctor evaluates the patients based on clinical practice.

Since this study is an observational study, the diagnosis and treatment process listed in the protocol is a clinically recommended process and is not mandatory. Treatment and clinical visit schedules for enrolled patients were determined by clinicians based on routine practice. This study collects patient information, including safety and efficacy data, based on routine diagnosis and treatment procedures. Although the protocol does not mandate clinical visits, physicians are encouraged to follow up patients who have not been seen for at least 6 months to collect treatment-related data and determine patient survival. Patients will be considered lost to follow-up if they have not been seen for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old; patients with metastatic NSCLC with at least one measurable brain metastases, the longest diameter of the brain metastases is 0.5 to 3 cm, and the brain metastases have not received radiotherapy; stable neurological symptoms and/or are receiving Corticosteroid therapy. In addition, the following conditions are raised:

1. Patients with negative driver-gene mutations who have not received systemic treatment before, and patients who have progressed after receiving neoadjuvant or adjuvant therapy, and the interval between disease progression or recurrence and the end of the last chemotherapy drug treatment is at least 6 months, and is allowed to enter this study;
2. Patients with known EGFR sensitive mutation, ALK rearrangement or ROS1 fusion must have received at least one EGFR or ALK, ROS1 fusion inhibitor treatment and had disease progression or drug intolerance.
3. Subjects with neurological symptoms can receive dexamethasone within 10 days before the first treatment, but the total daily dose is stable at no more than 4 mg or other Corticosteroids at the same dose. Subjects with neurologic symptoms but not receiving steroids should experience no seizures within 10 days prior to first treatment.

2. For patients with non-brain oligometastases, according to Response Evaluation Criteria in Solid Tumors Version 1.1 (mRECIST v1.1), there is at least 1 measurable or evaluable lesion in addition to brain metastases.

3. The Eastern Cooperative Oncology Group Physical Status Score (ECOG PS score) is 0-2 points.

4. The patient has a clear mind, can answer correctly, and has basically normal vision, etc., and can cooperate with cognitive function assessment 5. Expected survival time ≥ 12 weeks. 6. The patient has adequate organ and bone marrow functions, as defined below:

1. Blood routine: absolute neutrophil count ≥1.5×109/L; platelet count ≥100×109/L; hemoglobin content ≥9.0 g/dL.
2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); for patients with HCC, liver metastases, or a history/suspect of Gilbert syndrome (persistent or recurrent hyperbilirubinemia , mainly high unconjugated bilirubin, no evidence of hemolysis or liver disease), TBIL ≤ 3 × ULN; for patients without HCC and liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; for patients with HCC or with liver metastases, ALT or AST ≤ 5 × ULN.
3. Renal function: serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance (CCr) ≥ 50mL/min; urine test paper test results show urine protein <2+.
4. Coagulation function: activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5×ULN.

Exclusion Criteria:

1. Receive live attenuated vaccine within 4 weeks before enrollment or plan to receive live attenuated vaccine during the study.
2. Active, known or suspected autoimmune disease.
3. Known history of primary immunodeficiency.
4. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
5. Female patients who are pregnant or breastfeeding.
6. Untreated acute or chronic active hepatitis B or hepatitis C infection. Patients who are receiving antiviral treatment will be judged by doctors according to the individual conditions of the patients under the condition of monitoring the virus copy number.
7. History of dementia, Alzheimer's disease, Parkinson's disease and other diseases that can cause cognitive dysfunction
8. History of schizophrenia, severe anxiety, depression, or other mental illnesses
9. Uncontrolled concurrent diseases, including but not limited to:

   1. HIV-infected persons (HIV antibody positive).
   2. Serious infection that is active or poorly controlled clinically.
   3. Serious or uncontrolled systemic disease (such as severe mental, neurological disease, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, hepatic or renal disease, uncontrolled hypertension [i.e. Evidence of greater than or equal to CTCAE grade 2 hypertension after drug treatment]).
   4. Active bleeding or new thrombotic disease is taking therapeutic dose of anticoagulant drugs or bleeding tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC Patients With Symptomatic Brain Metastases
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial clinical benefit rate (CBR) | 6 months
Intracranial progression-free survival (PFS) | 1 year

SECONDARY OUTCOMES:
Intracranial objective response rate (ORR) | 1 year
Extracranial clinical benefit rate (CBR) | 1 year
Extracranial objective response rate (ORR) | 1 year
Extracranial progression-free survival (PFS) | 1 year
Clinical benefit rate (CBR) | 1 year
Objective response rate (ORR) | 1 year
Progression-free survival (PFS) | 1 year
Overall survival (OS) | 1 year
Incidence of neurological adverse events | 1 year
Incidence of severe adverse events | 1 year
Rate of decline in cognitive function | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No